CLINICAL TRIAL: NCT05526911
Title: A Phase 1, Drug-Drug Interaction Study to Evaluate the Safety, Tolerability, and the Induction Potential of TBAJ-876 on CYP3A4 and P-glycoprotein and the Inhibition Potential of TBAJ-876 on P-glycoprotein in Healthy Adult Subjects
Brief Title: A Phase 1, Drug-Drug Interaction Study of TBAJ-876 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBAJ-876-CL002
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Disease; Tuberculosis, Pulmonary; Tuberculosis; Multi Drug Resistant Tuberculosis; Drug Sensitive Tuberculosis; Drug-resistant Tuberculosis; Mycobacterium Tuberculosis Infection
Keywords: TBAJ-876; Diarylquinoline; DARQ
MeSH Terms: conditions — Lung Diseases; Tuberculosis, Pulmonary; Tuberculosis; Tuberculosis, Multidrug-Resistant | interventions — TBAJ-876; Midazolam; Digoxin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): The pharmacokinetics of midazolam, a CYP3A4 substrate, and digoxin, a P-gp substrate, will be studied before and after dosing with TBAJ-876.
  Interventions: Drug: TBAJ-876; Drug: Midazolam; Drug: Digoxin

INTERVENTIONS:
Drug: TBAJ-876 — * Day 6 to Day 13: 200 mg TBAJ-876 oral suspension, fed
  * Day 14 to Day 19: 165 mg TBAJ-876 oral suspension, fed
  * Day 20 and Day 21: 200 mg TBAJ-876 oral suspension, fasting
  * Day 22 to Day 24: 150 mg TBAJ-876 oral suspension, fed
Drug: Midazolam — Day 1 and Day 20: Midazolam oral syrup: 2 mg, fasted
Drug: Digoxin — Day 2 and Day 21: Digoxin tablet: 0.25 mg, fasted

SUMMARY:
A Phase 1, Drug-Drug Interaction Study to Evaluate the Safety, Tolerability, and the Induction Potential of TBAJ-876 on CYP3A4 and P-glycoprotein and the Inhibition Potential of TBAJ-876 on P-glycoprotein in Healthy Adult Subjects

DETAILED DESCRIPTION:
This study was a two-part, open-label drug-drug interaction study conducted in one study center in the United States. Two groups were planned, Group 1 and Group 2. Group 2 to be conducted based on the Group 1 results.

Group 1 to assess the induction potential of TBAJ-876 on the sensitive CYP3A4 substrate midazolam (M) and inhibition and induction potential of TBAJ-876 on the sensitive P-glycoprotein substrate Digoxin (D).

Group 2 was only to be conducted if the results of Group 1 show that TBAJ-876 is a moderate inducer of either CYP3A4 (geometric mean ratio [GMR] of midazolam area under the curve [AUC] <0.50 when co-administered with TBAJ-876) or P-glycoprotein (GMR of digoxin AUC <0.50 when co-administered with TBAJ-876) or a moderate inhibitor of P-glycoprotein (GMR of digoxin AUC ≥2.0 when co-administered with TBAJ-876). These results were used to decide that a second phase of the study was not needed.

If Group 1 concluded that TBAJ-876 is a moderate inducer or inhibitor, Group 2 had intended to quantify the magnitude of inhibition or induction of TBAJ-876 of the antiretroviral regimen TLD, a fixed dose combination of tenofovir disoproxil fumarate (TFD), lamivudine (3TC) and dolutegravir (DTG), a regimen likely to be used in future clinical studies of TBAJ-876 by subjects living with HIV

Safety was assessed throughout the study for all subjects. Safety assessments included physical examinations, vital signs, serial ECGs, adverse events (AEs), clinical and laboratory tests (including hematology, serum chemistry, coagulation, and urinalysis).

ELIGIBILITY:
Key Inclusion Criteria:

* Is a healthy adult male or female, 18 to 55 years of age (inclusive) at the time of screening.
* Has a body mass index (BMI) ≥18.5 and ≤32.0 (kg/m2) and a body weight of no less than 50.0 kg at the time of screening and check-in.
* Is medically healthy with no clinically significant screening results (e.g., laboratory profiles normal or up to Grade 1 per Division of Microbiology and Infectious Diseases (DMID) Toxicity Tables), as deemed by the Investigator.
* Has not used tobacco- or nicotine-containing products (including smoking cessation products), for a minimum of 6 months before dosing.
* Is willing and able to consume the entire high-calorie, high-fat breakfast meal in the timeframe required.

Key Exclusion Criteria:

* History or presence of significant cardiovascular abnormalities, heart murmur, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease as determined by the Investigator to be clinically relevant.
* Any musculoskeletal abnormality (severe tenderness with marked impairment of activity) or musculoskeletal toxicity (frank necrosis).
* Positive results at screening for Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HBsAg), or Hepatitis C antibodies (HCV).
* Positive Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) results within 6 days prior to Day 1.
* Current or history of prolonged QT syndrome.
* Family history of Long-QT Syndrome or sudden death without a preceding diagnosis of a condition that could be causative of sudden death (such as known coronary artery disease, congestive heart failure or terminal cancer).
* Use of any drugs or substances known to be inducers of CYP enzymes and/or P-gp, including St. John's Wort, within 30 days prior to the first dose of study drug.
* Is lactose intolerant.
* History or presence of allergic, or adverse response to midazolam, digoxin, dolutegravir, tenofovir, lamivudine or any related drugs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lombardi, MD, Study Chair — Global Alliance for TB Drug Development
Locations (1):
- TKL Research, Inc., Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 75 subjects were screened for the trial of whom 47 failed screening, 28 were randomized, and 26 completed treatment.
Pre-assignment Details: No participants were assigned to Group 2
Groups:
- Group 1: The pharmacokinetics of midazolam, a CYP3A4 substrate, and digoxin, a P-gp substrate, will be studied before and after dosing with TBAJ-876.
  TBAJ-876: • Day 6 to Day 13: 200 mg TBAJ-876 oral suspension, fed
  * Day 14 to Day 19: 165 mg TBAJ-876 oral suspension, fed
  * Day 20 and Day 21: 200 mg TBAJ-876 oral suspension, fasting
  * Day 22 to Day 24: 150 mg TBAJ-876 oral suspension, fed
  Midazolam: Day 1 and Day 20: Midazolam oral syrup: 2 mg, fasted
  Digoxin: Day 2 and Day 21: Digoxin tablet: 0.25 mg, fasted
Period: Overall Study
Arm/Group | Group 1
Started | 28
Completed | 26
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28
Height at Screening [Mean (Standard Deviation); unit: centimeters] | 167.3 (10.41)
Weight at Screening [Mean (Standard Deviation); unit: Kilogram] | 78.2 (19.86)
BMI at Screening [Mean (Standard Deviation); unit: kilogram per meter squared] | 28 (8.03)

OUTCOME MEASURES:

1. Primary Outcome: TBAJ-876 Effect on the Pharmacokinetics of the CYP-3A4 Substrate Midazolam in Healthy Adult Subjects: Pharmacokinetic Parameters AUC
Description: Geometric mean and range of midazolam's area under the (plasma concentration vs. time) curve when co-administered with TBAJ-876 versus when administered alone.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours; Day 20: pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours
Population: All participants enrolled in the study were included. Participants who were withdrawn prior to Day 20 are not included in the analysis with TBAJ-876. Participants were excluded from AUC 0-inf analysis if they did not have at least 3 observations presented along what appears to be a terminal elimination phase when individual subject plots of each analyte concentration vs time were inspected visually to identify log-linear terminal segments corresponding to an exponential elimination phase.
Measure: Geometric Mean (Full Range); unit: ng.hr/mL
Groups:
- Group 1: Midazolam
Arm/Group | Group 1
Number analyzed (Participants) | 28
ng.hr/mL
  Area under curve from time 0 hours to last quantifiable concentration (AUC 0-last), with TBAJ-876: number analyzed (Participants) | 26
  Area under curve from time 0 hours to last quantifiable concentration (AUC 0-last), with TBAJ-876 | 22.64 [7.98 to 43.78]
  AUC 0-last, alone | 25.22 [8.30 to 93.20]
  Area under the curve from time 0 hours to infinity (AUC 0-inf), with TBAJ-876: number analyzed (Participants) | 24
  Area under the curve from time 0 hours to infinity (AUC 0-inf), with TBAJ-876 | 24.28 [8.65 to 46.52]
  AUC 0-inf, alone: number analyzed (Participants) | 26
  AUC 0-inf, alone | 25.68 [8.79 to 98.22]

2. Primary Outcome: TBAJ-876 Effect on the Pharmacokinetics of the CYP-3A4 Substrate Midazolam in Healthy Adult Subjects: Pharmacokinetic Parameters CMAX
Description: Geometric mean and range of midazolam's maximum concentration when co-administered with TBAJ-876 versus when administered alone.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours; Day 20: pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours
Population: All participants enrolled in the study were included. Participants who were withdrawn prior to Day 20 are not included in the analysis with TBAJ-876.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Group 1
Number analyzed (Participants) | 28
ng/mL
  Maximum Concentration (Cmax), with TBAJ-876: number analyzed (Participants) | 26
  Maximum Concentration (Cmax), with TBAJ-876 | 7.26 [3.37 to 19.90]
  Cmax, alone | 8.90 [3.08 to 27.50]

3. Primary Outcome: TBAJ-876 Effect on the Pharmacokinetics of the CYP-3A4 Substrate Midazolam in Healthy Adult Subjects: Geometric Mean Ratios
Description: Geometric mean ratio of midazolam's area under the (plasma concentration vs. time) curve and Cmax when co-administered with TBAJ-876 versus when administered alone. Inference will be based on analysis of variance applied to log-transformed parameters.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours; Day 20: pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours
Population: All participants who completed the study were included. Participants were excluded from AUC 0-inf analysis if they did not have at least 3 observations presented along what appears to be a terminal elimination phase when individual subject plots of each analyte concentration vs time were inspected visually to identify log-linear terminal segments corresponding to an exponential elimination phase.
Measure: Geometric Mean (90% Confidence Interval); unit: ratio of geometric mean
Arm/Group | Group 1
Number analyzed (Participants) | 26
ratio of geometric mean
  AUC 0-last Ratio of geometric means of midazolam with TBAJ-876 to midazolam alone | 0.94 [.84 to 1.06]
  AUC 0-inf Ratio of geometric means of midazolam with TBAJ-876 to midazolam alone: number analyzed (Participants) | 23
  AUC 0-inf Ratio of geometric means of midazolam with TBAJ-876 to midazolam alone | 1 [.88 to 1.12]
  Cmax Ratio of geometric means of midazolam with TBAJ-876 to midazolam alone | .86 [.76 to .98]

4. Primary Outcome: TBAJ-876 Effect on the Pharmacokinetics of the P-gp Substrate Digoxin: Pharmacokinetic Parameters AUC
Description: Geometric mean of digoxin's area under the (plasma concentration vs. time) curve when co-administered with TBAJ-876 versus when administered alone, and similarly for the maximum concentration.
Time Frame: Day 2: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours; Day 21: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours
Population: as for outcome 3
Measure: Geometric Mean (Full Range); unit: ng.hr/mL
Arm/Group | Group 1
Number analyzed (Participants) | 26
ng.hr/mL
  AUC 0-last, with TBAJ-876 | 11.57 [0.03 to 33.24]
  AUC 0-last, alone | 7.64 [0.55 to 31.12]
  AUC 0-inf, with TBAJ-876: number analyzed (Participants) | 3
  AUC 0-inf, with TBAJ-876 | 24.57 [19.73 to 27.89]
  AUC 0-inf, alone: number analyzed (Participants) | 2
  AUC 0-inf, alone | 23.44 [19.86 to 27.67]

5. Primary Outcome: TBAJ-876 Effect on the Pharmacokinetics of the P-gp Substrate Digoxin: Pharmacokinetic Parameters CMAX
Description: Geometric mean of digoxin's Cmax when co-administered with TBAJ-876 versus when administered alone, and similarly for the maximum concentration.
Time Frame: as for outcome 4
Population: All participants who completed the study were included.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Group 1
Number analyzed (Participants) | 26
ng/mL
  Cmax, with TBAJ-876 | 1.19 [0.11 to 2.64]
  Cmax, alone | 1.01 [0.39 to 2.18]

6. Primary Outcome: TBAJ-876 Effect on the Pharmacokinetics of the P-gp Substrate Digoxin: Geometric Mean Ratio
Description: Geometric mean ratio of digoxin's area under the (plasma concentration vs. time) curve and Cmax when co-administered with TBAJ-876 versus when administered alone, and similarly for the maximum concentration. Inference will be based on analysis of variance applied to log-transformed parameters.
Time Frame: as for outcome 4
Population: All participants who completed the study were included.
Measure: Geometric Mean (90% Confidence Interval); unit: ratio of geometric mean
Arm/Group | Group 1
Number analyzed (Participants) | 26
ratio of geometric mean
  AUC 0-last Ratio of geometric means of digoxin with TBAJ-876 to digoxin alone | 1.51 [1.13 to 2.03]
  Cmax Ratio of geometric means of digoxin with TBAJ-876 to digoxin alone | 1.18 [.91 to 1.53]

7. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events (TEAE) in Group 1 Population
Description: Participants will be monitored for any adverse events from the signing of the consent form until the end-of-study visit. The Investigator or a Sub-Investigator will assess its relationship to the study drug.
  Note about ST segment elevation which was reported as a treatment-related adverse event. Upon review of the screening ECG, early repolarization was noted and therefore the ST segment elevation was considered pre-existing and not a TEAE however the AE remained in the database instead of being removed.
Time Frame: from date of the start of treatment to the end of study at 25 days
Population: Enrolled participants will be monitored for any adverse events from the signing of the consent form until the end-of-study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1
Number analyzed (Participants) | 28
Participants | 5

ADVERSE EVENTS:
Time Frame: Beginning of treatment on Day 1 through follow up on Day 32.
Description: Note about ST segment elevation which was reported as an adverse event (AE). Upon review of the screening ECG, early repolarization was noted and therefore the ST segment elevation was considered pre-existing and not an AE however the AE remained in the database instead of being removed.
Arm/Group | Group 1
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 9/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=28)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Oral discomfort (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Electrocardiogram PR interval elongation (Investigations) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Lethargy (Nervous system disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/11/NCT05526911/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT05526911/SAP_001.pdf